CLINICAL TRIAL: NCT01782248
Title: Self-consciousness in Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5289; 5289 (Other: HUS)
Record Dates: First submitted 2012-10-15; First posted 2013-02-01 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease; Fronto-temporal Lobar Dementia
MeSH Terms: conditions — Alzheimer Disease

ARMS (3):
- Alzheimer disease (Other): Patients with Alzheimer disease
  Interventions: Other: Questionnary and IRM
- Fronto-temporal lobar dementia (Other): Patients with Fronto-temporal lobar dementia
  Interventions: Other: Questionnary and IRM
- Control (Other): Control group
  Interventions: Other: Questionnary and IRM

INTERVENTIONS:
Other: Questionnary and IRM

SUMMARY:
The aim of this study is to characterize the deficit in critical components of personal identity (self-consciousness and social cognition) in patients with Alzheimer's disease (AD) and fronto-temporal lobar dementia (FTLD), compared to healthy elderly, combining a neuropsychology and multi-podal neuroimaging study.

We posit that the alteration of some aspects of self-consciousness (autobiographical memory, nosognosia, metacognition) and social cognition (theory of mind and facial) results in personality changes in the patients, primarily due to the alteration of self-consciousness in AD and to social cognition in FTLD.

ELIGIBILITY:
Inclusion Criteria:

* AD (McKhann et al, 1984 and Dubois et al, 2007) or FTLD (Neary et al, 1998 or Rascovsky et al, 2011)
* MMSE > or = 18
* Relative avaible

Exclusion Criteria:

* Contraindication to MRI
* Major depression
* Other central neurological condition

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2013-03-13 (Actual); Primary Completion 2022-03-12 (Estimated); Study Completion 2022-03-12 (Estimated)

PRIMARY OUTCOMES:
Characterize the deficit in critical components of personal identity in patients with Alzheimer's disease (AD) and fronto-temporal lobar dementia (FTLD), compared to healthy elderly, combining a neuropsychology and multi-podal neuroimaging study. | each month for 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France